CLINICAL TRIAL: NCT00135174
Title: Cost-Effectiveness of Routine Follow-up Visits in Patients With a Pacemaker: The FOLLOWPACE Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: College of Health Insurers/Society of Academic Hospitals, (Unknown); Dutch Working Group on Cardiac Pacing, (Unknown); Foundation Pacemaker Registry in The Netherlands, (Unknown)
Responsible Party: K.G.M. Moons, Julius Center for Health Sciences and Primary Care
Other Study IDs: CVZ/VAZ 01236
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Arrhythmia; Heart Diseases
Keywords: Pacemaker; routine; follow-up; complications; Quality of Life
MeSH Terms: conditions — Arrhythmias, Cardiac; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The overall objective of the study is to quantify the true prognostic value and cost-effectiveness of routine follow-up visits in patients who receive an approved pacemaker of any type for the first time.

DETAILED DESCRIPTION:
Specific objectives :

* To determine the incidence of complications occurring in the first year after implantation of a pacemaker.
* To determine the quality of life at one year after pacemaker implantation in comparison with the quality of life before implantation.
* To determine which baseline (patient and pacemaker related) characteristics measured during implantation are prognostic predictors for the occurrence of complications and quality of life after one year.
* To determine which characteristics measured during follow-up visits truly have added predictive value, and to what extent.
* To determine to what extent responsibilities for pacemaker check-up can be safely delegated to non-cardiologists (e.g. pacemaker technicians or manufacturers' delegates).

ELIGIBILITY:
Inclusion Criteria:

* Each patient aged 18 years or over receiving a pacemaker for the first time in one of the participating Dutch pacemaker implanting centers, is a potential candidate for the study.

Exclusion Criteria:

* Patients are not eligible if they refuse to sign informed consent on use of personal medical data.
* Patients who are taking any investigational (new) drug or have a non-approved or investigational pacemaker system which requires unusual follow-up regarding the pacemaker
* Patients having diseases that are likely to cause death or significant morbidity during the study period such as neoplasia and immune, infectious or degenerative diseases will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring a PM for conventional reasons.
Sampling Method: Non-Probability Sample
Enrollment: 1526 (Actual)
Dates: Start 2003-09; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Norbert van Hemel, M.D., Study Chair — University of Utrecht, Julius Center for Primary Care and Health Sciences; Karel G Moons, PhD, Study Chair — University of Utrecht, Julius Center for Primary Care and Health Sciences; Diederick E Grobbee, M.D., Study Chair — University of Utrecht, Julius Center for Primary Care and Health Sciences
Locations (1):
- Julius Center for Primary Care and Health Sciences, University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Udo EO, van Hemel NM, Zuithoff NP, Doevendans PA, Moons KG. Risk of heart failure- and cardiac death gradually increases with more right ventricular pacing. Int J Cardiol. 2015 Apr 15;185:95-100. doi: 10.1016/j.ijcard.2015.03.053. Epub 2015 Mar 5. PMID 25804349
- [Derived] Udo EO, van Hemel NM, Zuithoff NP, Doevendans PA, Moons KG. Prognosis of the bradycardia pacemaker recipient assessed at first implantation: a nationwide cohort study. Heart. 2013 Nov;99(21):1573-8. doi: 10.1136/heartjnl-2013-304445. Epub 2013 Aug 22. PMID 23969476
- [Derived] Udo EO, van Hemel NM, Zuithoff NP, Nijboer H, Taks W, Doevendans PA, Moons KG. Long term quality-of-life in patients with bradycardia pacemaker implantation. Int J Cardiol. 2013 Oct 3;168(3):2159-63. doi: 10.1016/j.ijcard.2013.01.253. Epub 2013 Feb 28. PMID 23453871
- [Derived] Udo EO, van Hemel NM, Zuithoff NP, Dijk WA, Hooijschuur CA, Doevendans PA, Moons KG. Pacemaker follow-up: are the latest guidelines in line with modern pacemaker practice? Europace. 2013 Feb;15(2):243-51. doi: 10.1093/europace/eus310. Epub 2012 Oct 24. PMID 23097223
- [Derived] Udo EO, van Hemel NM, Zuithoff NP, Kelder JC, Crommentuijn HA, Koopman-Verhagen AM, Voskuil T, Doevendans PA, Moons KG. Long-term outcome of cardiac pacing in octogenarians and nonagenarians. Europace. 2012 Apr;14(4):502-8. doi: 10.1093/europace/eur329. Epub 2011 Oct 23. PMID 22024601
- See also: Webpage with information on study center. — http://www.juliuscenter.nl
- See also: Electronic CRF pages and entire protocol can be viewed here. — http://www.followpace.nl